CLINICAL TRIAL: NCT04839029
Title: Bipolar Versus Monopolar Needlescopic En Bloc Transurethral Resection of Non-muscle Invasive Bladder Cancer: A Prospective Randomized Study
Brief Title: Bipolar Versus Mono-polar Needlescopic En Bloc TUR-BT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Waleed El-Shaer, MD, Associate professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDIRB2017122601-293
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Bladder Cancer; Bladder Neoplasm
Keywords: NMIBC; TURBT; En bloc resection
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bipolar En bloc TURBT (Experimental): patient subjected to bipolar Needlescopic En bloc resection of NMIBC
  Interventions: Procedure: Bipolar En bloc TURBT
- Monopolar En bloc TURBT (Active Comparator): patient subjected to Monopolar Needlescopic En bloc resection of NMIBC
  Interventions: Procedure: Monopolar En bloc TURBT

INTERVENTIONS:
Procedure: Bipolar En bloc TURBT — patients subjected to Bipolar resection of bladder tumor by Collins loop
  Arms: Bipolar En bloc TURBT
Procedure: Monopolar En bloc TURBT — patients subjected to Monopolar resection of bladder tumor by Collins loop (hot Knife)
  Arms: Monopolar En bloc TURBT

SUMMARY:
Non-muscle invasive bladder cancers (NMIBC) compose about 80% of bladder tumors. the stranded treatment of these tumors is TURBT.

en bloc resection of NMIBC yields better mascularis propria with better oncological outcomes

ELIGIBILITY:
Inclusion Criteria:

* confirmed primary NMIBC (Ta, Tis, T1)
* Age > 18 years

Exclusion Criteria:

* MIBC
* anterior located mass ( difficult or non visualized)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Quality of tumor Resection | immediatly post operative
  presence of detrusor muscle
adequacy of tumor Resection | 2 to 6 weeks postoprative
  Presence of residual tumor at the bed of previously resected NMIBC

SECONDARY OUTCOMES:
Complications | within 30 days post-operative
  Modified Clavien-Dindo classification scale

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-Shaer, M.D, Principal Investigator — Faculty of medicine, Banha university
Locations (1):
- Banha university hospital, Banhā, Qalyubia Governorate, Egypt